CLINICAL TRIAL: NCT06389500
Title: Hepatic Arterial Infusion Chemotherapy Combined With Adebrelimab and Lenvatinib for Conversion Treatment of Potentially Resectable, Locally Advanced Biliary Tract Cancer: a Single-arm, Exploratory Clinical Study
Brief Title: HAIC+Adebrelimab+Lenvatinib for Conversion Treatment of Potentially Resectable, Locally Advanced Biliary Tract Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Harbin Medical University (Other)
Responsible Party: Principal Investigator, Yubao Zhang, MD, Harbin Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1316-HLJ-006
Record Dates: First submitted 2024-04-24; First posted 2024-04-29 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Biliary Tract Cancer
Keywords: Adebrelimab; Hepatic Arterial Infusion Chemotherapy; Lenvatinib; Potentially Resectable Biliary Tract Cancer
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HAIC+Immune-targeted therapy (Experimental): Hepatic arterial infusion chemotherapy combined with adebrelimab and lenvatinib
  Interventions: Drug: Adebrelimab; Drug: Lenvatinib; Procedure: Hepatic Arterial Infusion Chemotherapy

INTERVENTIONS:
Drug: Adebrelimab — Adebrelimab, IV
  Other Names: SHR-1316
Drug: Lenvatinib — Lenvatinib, PO
  Other Names: Lenvatinib Mesilate Capsules
Procedure: Hepatic Arterial Infusion Chemotherapy — GC regimen±5-FU

SUMMARY:
This is a single-arm, exploratory, phase II trial to evaluate the efficacy and safety of hepatic arterial infusion chemotherapy combined with adebrelimab and lenvatinib for borderline resectable, locally advanced biliary tract cancer.

DETAILED DESCRIPTION:
This study plans to recruit 30 patients with borderline resectable, locally advanced biliary tract cancer who have not received treatment， abserve and evaluate the efficacy and safety of hepatic arterial infusion chemotherapy combined with adebrelimab and lenvatinib.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 to 75 years old, male or female;
2. Biliary tract malignant tumors confirmed by histology or cytology, with measurable tumor lesions (spiral CT or MR scan ≥10mm, meeting RECIST 1.1 standards);
3. Borderline resectable, locally advanced biliary malignant tumors, including gallbladder cancer, intrahepatic cholangiocarcinoma, hilar cholangiocarcinoma, and distal cholangiocarcinoma;
4. Clinical stage: gallbladder cancer stage: IIIA-IVB; intrahepatic cholangiocarcinoma stage: IIA-IV; hilar cholangiocarcinoma stage: IIIB-IVB; distal cholangiocarcinoma stage: IIIA-IV;
5. Expected survival > 3 months;
6. ECOG PS score: 0-1 points;
7. Liver function classification is Child-Pugh ≤7;
8. Never received prior systemic treatment for biliary tract tumors;
9. No peritoneal metastasis or other distant metastasis;
10. Normal function of major organs;
11. Women of childbearing age must have a negative pregnancy test (βHCG) before starting treatment, and women of childbearing potential and men (who have sexual active with women of childbearing potential) must agree to effective contraception uninterrupted for the duration of the treatment and for 6 months after the last therapeutic dose;
12. Patients voluntarily enrolled in the study by signing an informed consent form.

Exclusion Criteria:

1. Patients diagnosed with periampullary cancer;
2. Previous or concurrent other malignant tumours within 5 years, except cervical carcinoma in situ, cutaneous squamous cell carcinoma or basal cell carcinoma of the skin that has been basically controlled;
3. Those with uncontrolled, symptomatic brain metastases or a history of uncontrollable mental illness or severe intellectual or cognitive dysfunction;
4. Pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonitis, drug-related pneumonia and severely impaired lung function;
5. Suffering from active autoimmune diseases, history of autoimmune diseases, such as interstitial pneumonia, colitis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism; Reduced thyroid function after thyroid hormone replacement therapy can be included;
6. Have a history of immunodeficiency, including testing positive for HIV, suffering from other acquired or congenital immunodeficiency diseases, or a history of organ transplantation and allogeneic bone marrow transplantation;
7. Subjects have cardiovascular clinical symptoms or diseases that cannot be well controlled, including but not limited to: 1) NYHA class II or above heart failure; 2) Unstable angina; 3) Myocardial infarction within 1 year; 4) Clinically significant supraventricular or ventricular arrhythmia requiring clinical intervention;
8. Severe active infection requiring intravenous antibiotic treatment occurs during the screening period;
9. Those who are allergic to experimental drugs;
10. Patients who cannot comply with the trial protocol or cannot cooperate with follow-up visits;
11. Those who the researcher believes are not suitable to participate in this trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2027-05-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
R0 resection rate | up to 24 months
  Postoperative staining results showed that the lesion was completely resected, and pathological biopsy of the transverse and longitudinal margins were negative.
Surgery conversion rate | up to 24 months
  Proportion of patients who can undergo surgical resection among all enrolled patients

SECONDARY OUTCOMES:
Objective response rate | up to 24 months
  The proportion of patients whose tumor volume shrinks to a predetermined value and can maintain the minimum time limit, which is the sum of the proportions of complete remission and partial remission.
pathological complete response rate | up to 24 months
  After preoperative treatment and surgery, there are no residual viable tumor cells in the tumor bed in the postoperative specimen (%RVT=0)
Major pathological response rate | up to 24 months
  After preoperative treatment and surgery, the proportion of residual viable tumor cells in the tumor bed in the postoperative specimen is less than or equal to 10% (%RVT≤10)*
Recurrence-free survival | up to 24 months
  Duration from surgical resection to first recurrence or death from any cause
Overall survival | up to 24 months
  Overall survival is measured from the first dose of study drug until death from any cause.
AEs | up to 24 months
  Incidence, nature, and severity of adverse events graded according to the NCI CTCAE v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Yubao Zhang, MD, Principal Investigator — Harbin Medical University Affiliated Cancer Hospital

IPD SHARING:
Plan to Share IPD: No